CLINICAL TRIAL: NCT00002223
Title: Ritonavir (ABT-538)/Indinavir Combination Treatment in HIV-Infected Patients Previously Receiving Indinavir 800 mg TID
Brief Title: A Study of Ritonavir/Indinavir Combination in HIV-Infected Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott (Industry)
Purpose: Treatment
Other Study IDs: 245E; M98-823
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2009-02-20 (Estimated); Status verified 2009-02

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Adolescent Behavior; HIV Protease Inhibitors; Ritonavir; Indinavir
MeSH Terms: conditions — HIV Infections; Adolescent Behavior | interventions — Indinavir; Ritonavir

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Ritonavir

SUMMARY:
The purpose of this study is to determine how many HIV-infected patients continue taking ritonavir/indinavir combination after having taken indinavir three times a day as part of their anti-HIV drug therapy. This study also examines the safety and effectiveness of the ritonavir/indinavir combination.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV infection.
* CD4 cell count greater than 100 cells/microliter.
* HIV RNA levels greater than 400 copies/microliter using the Roche Ultrasensitive assay.
* No acute illness.
* Consent of parent or guardian if less than legal age.
* No prior enrollment in this study.
* All entry criteria for this study met within 15 days prior to enrollment.

Exclusion Criteria

Co-existing Condition:

Patients with any of the following symptoms or conditions are excluded:

Any condition that in the opinion of the investigator may obscure proper observation of the safety or activity of the treatment regimens used in this study.

Concurrent Medication:

Excluded:

* Concurrent non-nucleoside reverse transcriptase inhibitors as part of the antiretroviral regimen.
* Any of the following medications with ritonavir:
* midazolam, clorazepate, diazepam, estazolam, flurazepam, triazolam, zolpidem, quinidine, amiodarone, encainide, flecainide, propafenone, bepridil, terfenadine, astemizole, cisapride, bupropion, clozapine, rifabutin, meperidine, propoxyphene, piroxicam, pimozide, dihydroergotamine, and ergotamine.
* Any of the following medications with indinavir:
* terfenadine, astemizole, cisapride, triazolam, midazolam. No requirement for rifampin or ketoconazole.
* Any concurrent treatment with other protease inhibitors.
* Other concurrent medication (including over-the-counter medicine or alcohol) without the knowledge and permission of the primary investigator.

Patients with the following prior conditions are excluded:

* History of significant drug hypersensitivity.
* Psychiatric illness that precludes compliance with the protocol.
* Receipt of investigational drug within 30 days prior to administration of study drug.
* History of acute or chronic pancreatitis.
* Anticipation of poor patient compliance with protocol.

Prior Medication:

Excluded:

Prior treatment with ritonavir.

Risk Behavior:

Excluded:

History of active substance abuse (i.e., recreational drugs or alcohol).

Included:

- Indinavir 800 mg three times a day plus unspecified nucleosides for at least 3 months.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - AIDS Healthcare Foundation, Los Angeles, California
  - Tower Infectious Diseases, Los Angeles, California
  - Urgent Care Ctr / North Broward Hosp District, Fort Lauderdale, Florida
  - Goodgame Med Ctr / Central Florida Research Initiati, Maitland, Florida
  - Mount Sinai Med Ctr, New York, New York
  - Stephen Hauptman, Philadelphia, Pennsylvania